CLINICAL TRIAL: NCT03035578
Title: Development of a Morphine Pharmacokinetic and Pharmacodynamic Model for the Neonatal Population
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: research project has been abandoned primarily because of the excessive delays associated with past challenges in obtaining approval from Health Canada
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrew James, Interim Head, Division of Neonatology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1000053067
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pain; Drug Effect
Keywords: Pharmacokinetics; Pharmacodynamics; Morphine; Neonatal
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphine Blood and Saliva sampling (Experimental): The infants will receive a 50 mcg/kg loading dose of morphine followed by a constant infusion.Morphine Injection: 10mg/mL, 1mL ampoules.Two strengths of stock syringes:
  a)patients <1.5kg, morphine 0.5mg/25mL; b)patients 1.5kg to <5kg, morphine 1mg/25mL.
  Time blood samples will be collected for measurement of whole blood concentration of morphine in 24h. Total morphine, morphine-3-glucuronide and morphine-6-glucuronide concentrations; volume of blood required is 0.25 ml. Sparse sampling strategy will be used for those neonates < 1250; total volume of blood required is 0.50 ml. Frequent sampling strategy will be used for those neonates ≥ 1250 gm; total volume of blood required is 0.50 ml.Saliva samples will be collected at 10 and 30 minutes and at 6, 12 and 24h after morphine infusion started.100 uL of saliva, captured using a collection swab.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Sampling blood for development of Morphine Pharmacokinetic/Pharmacodynamic Model for Neonatal Population
Drug: Morphine — Sampling saliva for development of Morphine Pharmacokinetic/Pharmacodynamic Model for Neonatal Population

SUMMARY:
This research aims to study what the baby's body does with morphine and how morphine works in the baby's body. One hundred newborn babies will be enrolled in this study. With a better understanding of the drug doctors and nurses will have more information and better administer the drug in case of pain, stress or discomfort.

DETAILED DESCRIPTION:
Critically ill immature preterm infants experience multiple noxious stimuli while receiving care in the Neonatal Intensive Care Unit (NICU). These noxious stimuli include, but are not limited to: venipuncture; insertion of intravenous and arterial catheters; suctioning of the nose, mouth and oropharynx; endotracheal intubation for mechanical ventilation; insertion of chest drains; repositioning and other types of patient manipulation. The delivery of optimal doses of analgesics for these noxious stimuli is a major challenge due to the lack of knowledge about drug disposition and its effects in this patient population.

Morphine is the commonest analgesic used in the NICU. The Premature Infant Pain Profile (PIPP) is used to quantify pain in the NICU1. This objective score, which combines physiological and behavioural variables defining levels of discomfort, is used as a guide for the use of morphine in newborn infants. Multidimensional pain assessment tools, such as PIPP, can easily identify behaviour in healthy infants undergoing painful events, however, its efficiency is questionable when applicable to critically ill premature infants with neurological impairment, where the pain processing and modulation may be altered. Pharmacokinetics/Pharmacodynamics (PKPD) models can be used to quantitatively describe and predict drug disposition in the blood and the target organ (e.g., brain) in relation to doses and patient characteristics. Although there has been a global effort to describe morphine plasma levels in this population using a pharmacokinetic modelling approach2-5, PKPD model development has not been reported. The study of morphine pharmacokinetics to determine the optimal dose for balancing analgesia/sedation together with the design of pharmacodynamic model for morphine may provide a better understanding of nociception/pain profile based on the physiological variables of immature infants. Moreover, the PKPD model may be used to achieve optimal therapeutic effects through individualised model-based dose selection. Objective: This study is composed by four main objectives:

1. First: Define target morphine plasma and brain concentrations. To this end, we will develop a morphine PKPD model based on population PK characteristics and morphine effects captured by functional readout of central nervous system function;
2. Second: Develop an opportunistic sampling method for fragile populations based on saliva sampling;
3. Third: Compare pharmacokinetic parameters calculated from saliva with plasma sample;
4. Fourth: Application of the morphine PKPD model for prediction of optimal morphine dosing in individual patients using the Bayesian framework of model refinement.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 24 completed weeks.
* Clinically prescribed to commence a continuous morphine infusion.

Exclusion Criteria:

* Gestational age < 24 completed weeks.
* Critically ill infant unlikely to survive for more than 72 hours.
* Prolonged fetal exposure to morphine, any other narcotic, or methadone, as a consequence of maternal use of the drug.
* Any postnatal exposure to morphine during the 72 hours prior to the commencement of the second morphine infusion.
* Neonates with impaired cardiac, hepatic or renal functioning as defined by clinical signs of impaired perfusion, abnormal liver function tests, or an elevated serum creatinine.
* Neonates with seizures.
* The attending neonatologist considers that participation in the study is contraindicated.

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Target Morphine Plasma Concentration | 12 months (blood sampling and modeling)
  Sparse sampling coupled with population (mixed effects) method will be used to design the morphine pharmacokinetics phase. This method captures pharmacokinetics data from many subjects (learning about population), which are based on a relatively few number of samples per patient (learning about individual characteristics considering the large number of samples).Population pharmacokinetic parameters will be estimated using a non-linear mixed effects modelling with NONMEM software.

SECONDARY OUTCOMES:
Brain Morphine Concentrations | 12 months (a-eeg collection and modeling)
  The drug effect will be design using the sigmoid modelling. The effect of drugs modeled by relating drug effect to the drug concentration (obtain in the primary outcome). The pain scores and amplitude-integrated electroencephalography (aEEG) will be used as markers of drug effect on the central nervous system for the development of the pharmacodynamic model. The effect-site concentration will be validated by comparing the predicted time of peak effect with the time of peak effect of aEEG effect. Heart rate, respiratory rate, blood oxygen saturation, and blood pressure will be captured continuously through neonatal computational platform with the intent to investigate, other pharmacodynamic relationship using the sigmoid modelling.

IPD SHARING:
Plan to Share IPD: No